CLINICAL TRIAL: NCT00182520
Title: A Study of Topiramate Augmentation in Serotonin Reuptake Inhibitor (SRI) -Refractory Obsessive Compulsive Disorder
Brief Title: Efficacy of Adding Topiramate to Current Treatment in Refractory Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Janssen-Ortho Inc., Canada (Industry); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-133
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Treatment Refractory Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Topiramate
  Interventions: Drug: Topiramate
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Topiramate — 25 mg - 400 mg/day x 12 weeks
  Other Names: Topomax
  Arms: 1
Drug: placebo — 25 - 400 mg/day x 12 weeks
  Arms: 2

SUMMARY:
SRI's are considered first-line treatments for OCD, however many patients continue to have significant symptoms despite an adequate trial of an SRI. Neuroimaging studies have shown that the glutamate neurological system is involved in OCD. This study will test the safety and efficacy of topiramate, a drug, which targets glutamate, in the treatment of OCD, where the OCD has been un-responsive, or partially responsive to regular SRI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with primary DSM- IV OCD
* Completion of a 14-week open label trial of one the following SRI's: fluoxetine 80 mg/day, paroxetine 60 mg/day, fluvoxamine 300 mg/day, clomipramine 250 mg/day, sertraline 200 mg/day, citalopram 60 mg/day, escitalopram 30 mg/day and demonstrating a non or partial responses to SRI treatment (CGI-I of 3 or 4, Y-BOCS reduction of < 35%)
* Stable (8 wks or longer) concurrent medications including benzodiazepines, sedative hypnotics, antipsychotics, and antidepressants.

Exclusion Criteria:

* Any other primary DSM-IV diagnosis; DSM-IV criteria for body dysmorphic disorder, bipolar affective disorder, schizophrenia, psychotic disorder, current alcohol/substance abuse.
* A previous adequate trial of topiramate
* Comorbid major depressive disorder diagnosis which predates OCD diagnosis
* Cognitive behavioural therapy or additional psychotherapy in past four months
* Allergy or hypersensitivity to topiramate
* BMI < 20
* History of kidney stones

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-01; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 12 weeks
Clinical Global Impression - Improvement ≤ 2 | 12 weeks

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | 12 weeks
Sheehan Disability Scale | 12 weeks
Beck Depression Inventory | 12 weeks
PI-SWUR Hoarding Scale | 12 weeks
Self Report Y-BOCS | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael VanAmeringen, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada